CLINICAL TRIAL: NCT01799915
Title: Natural History Study of Synucleinopathies
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 08-1408
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Patients With Synucleinopathies; Neurogenic Orthostatic Hypotension; Pure Autonomic Failure; REM Sleep Behavior Disorder; Parkinson Disease; Dementia With Lewy Bodies; Multiple System Atrophy; Shy-Drager Disease
MeSH Terms: conditions — Pure Autonomic Failure; REM Sleep Behavior Disorder; Parkinson Disease; Lewy Body Disease; Multiple System Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Sample for DNA processing
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- REM sleep behavior disorder, RBD: Patients that have rapid eye movement sleep behavior disorder.
- multiple system atrophy: is a neurodegenerative disorder charaterized by abnormal alpha-synuclein deposition in the cytoplasm of oligodendroglial cells in the CNS, and typically sparing peripheral autonomic nerves.
- Pure Autonomic failure: A neurodegenerative disorder characterized by loss of peripheral noradrenergic fibers, with low levels of plasma norepinephine.
- Parkinson disease: A degenerative disorder of the central nervous system that leads to termors, difficulty walking, movement and coordination.
- Dementia with Lewy bodies: A neurodegenerative disorder similar to PAF and PD with the accumulation of Alpha-synuclein in the CNS however DLB patients develop dementia.

SUMMARY:
Synucleinopathies are a group of rare diseases associated with worsening neurological deficits and the abnormal accumulation of the protein α-synuclein in the nervous system. Onset is usually in late adulthood at age 50 or older. Usually, synucleinopathies present clinically with slowness of movement, coordination difficulties or mild cognitive impairment. Development of these features indicates that abnormal alpha-synuclein deposits have destroyed key areas of the brain involved in the control of movement or cognition. Patients with synucleinopathies and signs of CNS-deficits are frequently diagnosed with Parkinson disease (PD), dementia with Lewy bodies (DLB) or multiple system atrophy (MSA).

However, accumulation of alpha-synuclein and death of nerve cells can also begin outside the brain in the autonomic nerves. In such cases, syncucleinopathies present first with symptoms of autonomic impairment (unexplained constipation, urinary difficulties, and sexual dysfunction). In rare cases, hypotension on standing (a disorder known as orthostatic hypotension) may be the only clinical finding. This "pre-motor" autonomic stage suggests that the disease process may not yet have spread to the brain.

After a variable period of time, but usually within 5-years, most patients with abnormally low blood pressure on standing develop cognitive or motor abnormalities. This stepwise evolution indicates that the disease spreads from the body to the brain. Another indication of this spread is that acting out dreams (i.e., REM sleep behavior disorder, RBD) a problem that occurs when the lower part of the brain is affected, may also be the first noticeable sign of Parkinson disease.

The purpose of this study is to document the clinical features and biological markers of patients with synucleinopathies and better understand how these disorders evolve over time. The study will involve following patients diagnosed with a synucleinopathy (PD/DLB and MSA) and those believed to be in the "pre-motor" stage (with isolated autonomic impairment and/or RBD). Through a careful series of follow-up visits to participating Centers, we will focus on finding biological clues that predict which patients will develop motor/cognitive problems and which ones have the resilience to keep the disease at bay preventing spread to the brain. We will also define the natural history of MSA - the most aggressive of the synucleinopathies.

DETAILED DESCRIPTION:
α-synuclein is a small protein of 140 amino acids that is highly expressed in the brain. It's function remains poorly understood.10 Synucleinopathies are a group of neurodegenerative diseases associated with the abnormal accumulation of α-synuclein within cytoplasmic inclusions in neurons or oligodendroglia. These α-synuclein containing cytoplasmic aggregates occur throughout the brain, producing cell death and specific motor, autonomic and cognitive dysfunction in four phenotypically distinct synucleinopathies. When α-synuclein deposition occurs in neurons it aggregates into Lewy bodies, producing Parkinson disease (PD), dementia with Lewy bodies (DLB) or pure autonomic failure (PAF). Whereas in multiple system atrophy (MSA) neuronal death probably occurs as a consequence of α-synuclein aggregation in oligodendroglia.

A characteristic feature of the synucleinopathies is that they can all begin with varying degrees of autonomic dysfunction as the sole clinical feature - implying an initial diagnosis of isolated (pure) autonomic failure 11. After a variable period of time, but usually less than 5 years, only a small number of patients remain with a pure autonomic failure phenotype, but careful follow-up is lacking 11. Most patients develop cognitive or motor abnormalities (or both) and the patient is then diagnosed with PD, DLB or MSA.

This stepwise clinical progression suggests that the neurodegenerative process can in rare cases remain confined to autonomic neurons12, but more frequently spreads to affect additional areas of the central nervous system (CNS). This unique feature of the synucleinopathies poses diagnostic challenges and potential therapeutic opportunities.

The challenges are first, to determine whether PAF is a distinct disease or is always a prodromal phase of PD, DLB or MSA and second, to discover biomarkers that predict spread to motor and cognitive neurons. Such biomarkers would allow testing of disease-modifying strategies to delay or stop the neurodegenerative process in the pre-motor or pre-dementia phase. Aim 2 will focus on defining the natural history of MSA, the most aggressive of the synucleinopathies. This prospective observational study will establish disease-specific milestones for use in future clinical trials.

Obstacles to identifying biomarkers predicting further CNS involvement are that most medical centers only see patients with synucleinopathies when they already have developed motor and cognitive involvement, and that PAF and MSA are rare disorders. In this context the Autonomic Disorders Consortium (ADC) within the Rare Diseases Clinical Research Network (RDCRN) of the National Institutes of Health (NIH) was created with the objective of providing a better understanding of the variability, progression, and natural history of neurodegenerative synucleinopathies. Continuing this observational study, and increasing its power by including additional academic centers from the U.S., South America, and Europe, will allow us to define the natural history of these diseases and establish the sensitivity and specificity of the proposed biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female patients will be included
2. Aged 18 or over
3. Referred to any of the participating consortium sites with orthostatic intolerance, defined as symptoms of dizziness or lightheadedness in the standing position that disappear when supine.

Exclusion Criteria:

1. Diabetes according to the American Diabetes Association criteria
2. Congestive heart failure
3. Lupus or other collagen vascular disease
4. Systemic illness thought to be responsible for the orthostatic intolerance
5. Drug-induced orthostatic hypotension (i.e., the use of alpha-blockers, diuretics, tricyclic antidepressants or others thought by the investigator to play an important role in the patient's orthostatic hypotension)
6. Isolated vasovagal syncope
7. Inability to comply with the protocol, e.g. uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary autonomic disorders are a group of diseases that usually begin in adulthood with the inability to stand because of dizziness, lightheadedness and fainting. Symptoms are the result of a dysfunction in the autonomic nerves that regulate blood pressure and heart rate, and are either related to the accumulation of abnormal protein deposits and a primary neurodegenerative process (like Parkinson's disease, pure autonomic failure, dementia with Lewy bodies and multiple system atrophy), secondary to genetic abnormalities (dopamine-beta-hydroxylase deficiency), an autoimmune process (autoimmune ganglionopathy), or because of a direct injury to the nerves involved in buffering blood pressure fluctuations (acquired baroreflex failure).
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2011-06 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
To create a database of primary autonomic disorders that will serve as a phenotyping core. | 5 years
  We will create an enrollment database of patients with primary autonomic disorders. All patients will have standardized phenotyping evaluations that will combine clinical, physiological and biochemical strategies to characterize complex autonomic phenotypes, both known and still undiscovered.

SECONDARY OUTCOMES:
To define the natural history of neurogenic orthostatic hypotension and identify predictive biomarkers of autonomic disorders | 5 years
  We will map the natural history of primary autonomic failure and test the hypothesis that pure autonomic failure (PAF) is a neurodegenerative synucleinopathy that remains confined to the autonomic nervous system. We will also identify biomarkers that can distinguish patients with PAF from those with early (i.e., "pre-motor") MSA, PD, DLB or autonomic failure as a result of another disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Horacio C Kaufmann, MD, Principal Investigator — NYU MEDICAL CENTER
Locations (8):
- United States (5):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - NYU Medical Center, New York, New York
  - Vanderbilt Univeristy, Nashville, Tennessee
- FLENI - Fundación para la Lucha contras las Enfermedades Neurológicas, Buenos Aires, Argentina
- Seoul National University Hospital, Seoul, South Korea
- BioCruces Research Institute - Hospital Universitario de Cruces, Bilbao, Spain

REFERENCES:
- [Derived] Palma JA, Vernetti PM, Perez MA, Krismer F, Seppi K, Fanciulli A, Singer W, Low P, Biaggioni I, Norcliffe-Kaufmann L, Pellecchia MT, Marti MJ, Kim HJ, Merello M, Stankovic I, Poewe W, Betensky R, Wenning G, Kaufmann H. Limitations of the Unified Multiple System Atrophy Rating Scale as outcome measure for clinical trials and a roadmap for improvement. Clin Auton Res. 2021 Apr;31(2):157-164. doi: 10.1007/s10286-021-00782-w. Epub 2021 Feb 7. PMID 33554315
- [Derived] Norcliffe-Kaufmann L, Kaufmann H, Palma JA, Shibao CA, Biaggioni I, Peltier AC, Singer W, Low PA, Goldstein DS, Gibbons CH, Freeman R, Robertson D; Autonomic Disorders Consortium. Orthostatic heart rate changes in patients with autonomic failure caused by neurodegenerative synucleinopathies. Ann Neurol. 2018 Mar;83(3):522-531. doi: 10.1002/ana.25170. Epub 2018 Mar 10. PMID 29405350